CLINICAL TRIAL: NCT07180537
Title: Transforming Health Habits: Evaluating an Online Wellness Program for Individuals With Rheumatological Conditions
Brief Title: Creating Health Course Study for People With Rheumatological Conditions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Terry L. Wahls (Other)
Responsible Party: Sponsor-Investigator, Terry L. Wahls, Clinical Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 202503591
Record Dates: First submitted 2025-09-04; First posted 2025-09-18 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Rheumatoid Arthritis; Sjogren's Syndrome; Systemic Lupus Erythematosus; Mixed Connective Tissue Disease; Psoriatic Arthritis
Keywords: diet; self-care; internet course
MeSH Terms: conditions — Arthritis, Rheumatoid; Sjogren's Syndrome; Lupus Erythematosus, Systemic; Mixed Connective Tissue Disease; Arthritis, Psoriatic

STUDY DESIGN:
Intervention Model Description: waitlist control
Who Masked: Investigator
Masking Description: Investigator will be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention: Creating Health Online course (Experimental): This arm will begin the intervention immediately after randomization
  Interventions: Behavioral: Creating Health Online Course
- Delayed Intervention: Creating Health Online course (Other): This is the control arm.
  Interventions: Behavioral: Delayed access to Creating Health Online Course

INTERVENTIONS:
Behavioral: Creating Health Online Course — Immediate access to an online audio and video course with education about strategies to grow and improve resilience, diet quality, exercise, stress reduction and self-care
  Other Names: Online wellness course
  Arms: Immediate Intervention: Creating Health Online course
Behavioral: Delayed access to Creating Health Online Course — Delayed access (12-week delay) to an online audio and video course with education about strategies to grow and improve resilience, diet quality, exercise, stress reduction and self-care
  Other Names: Online wellness course
  Arms: Delayed Intervention: Creating Health Online course

SUMMARY:
The goal of this project is to critically evaluate the effectiveness of an online health program designed to improve diet and self-care in patients with rheumatological conditions, including rheumatoid arthritis (RA), Sjogren's syndrome (SS), systemic lupus erythematosus (SLE), mixed connective tissue disease (MCTD), psoriatic arthritis (PsA), Additionally, investigators will assess the program's effectiveness, as well as the challenges and facilitators involved in using an online wellness program to reduce fatigue and enhance the quality of life in patients suffering from these conditions.

DETAILED DESCRIPTION:
The goal of this project is to critically evaluate the effectiveness of an online health program designed to improve diet and self-care in patients with rheumatological conditions, including rheumatoid arthritis (RA), Sjogren's syndrome (SS), systemic lupus erythematosus (SLE), mixed connective tissue disease (MCTD), psoriatic arthritis (PsA),. Additionally, we will assess the program's effectiveness, as well as the challenges and facilitators involved in using an online wellness program to reduce fatigue and enhance the quality of life in patients suffering from these conditions.

Once the eligibility criteria are established and consent is obtained, investigators will invite study participants randomized to the intervention arm to the online course via email. Participants will be required to create a password to access the course. The online course and supplementary resources will be hosted on a secure website through the UIowa Canvas Classroom platform. Participants will progress through the online health course modules similarly to a non-graded online course. Within the course, there are exercises and personal assessments designed to enhance the participants' experience and success.

The course will cover various topics, including modules on developing an inner game plan, a food intervention plan, a physical intervention plan, and an increased resilience plan. The fourth module will propose various strategies to improve health beyond diet and exercise, such as the use of supplements, light therapy, detoxification, improved sleep, stress reduction, and other strategies to enhance bodily resilience.

Participants are encouraged to communicate and collaborate with their healthcare teams to personalize their treatment and determine whether the strategies suggested in the course are appropriate for their individual healthcare needs. This study aims to provide dietary education to a broader sample size than previously studied, including patients with limited resources such as financial constraints and geographic barriers that restrict access to registered dietitians experienced in dietary instruction for various rheumatological conditions. There is a growing interest in delivering education and support through an online platform to improve diet quality and self-care practices for autoimmune patients.

This study will utilize a randomized single-blind waitlist control design to evaluate the impact of the online course, which includes materials covering a modified Paleolithic elimination (MPE) diet, nutrient-dense vegetarian diets, Mediterranean diets, stress reduction techniques, and exercise strategies designed for autoimmune patients. Data will be collected in the short term (after 3 months) and long term (at the end of 6 months) to analyze the effects of the online wellness program on quality of life (QoL) and related outcomes among individuals with RA, SS, SLE, MCTD, PsA.

Investigators will request that study participants complete their baseline assessments within approximately 7 to 14 days following consent. Participants will receive an individual link to their baseline assessments via REDCap. Patients will be randomized into different study arms based on their baseline fatigue severity scores.

The proposed study will be conducted entirely online. The schedule will include three virtual visits at three-month intervals (months 0, 3, and 6). Online questionnaires will be distributed via REDCap to assess fatigue, quality of life, and dietary information according to the study schedule (months 0, 3, and 6).

ELIGIBILITY:
Inclusion criteria:

1. A diagnosis of one of the following: Rheumatoid Arthritis (RA), Sjogren's Syndrome, Systemic lupus erythematosus (SLE), Mixed connective tissue disease (MCTD), or Psoriatic Arthritis (PsA), as documented by their treating specialist or primary care provider, as reported by the participant.
2. Must be age 18 and older, at time of consent.
3. Must be fluent in both speaking and reading English.

   *Study participant must be able to read and comprehend informed consent document and speak with study staff about study document content. Study staff will use discretion in determining whether the study participant can clearly communicate with staff and comprehend the study material during the consent call or prior to the call.
4. Must have access to high-speed internet with devices capable of audio/video streaming.
5. Must be willing to participate in an online health course designed to improve dietary intake and self-care routines to help improve cellular function and health, and complete online surveys over the course of a 6-month period.
6. Individuals must pass the Short Portable Mental Status Questionnaire with scores for normal mental functioning (up to 2 errors). Cognitive impairment as measured by the SPMS Questionnaire could interfere with the completion of the online course.

SCORING* 0-2 errors: normal mental functioning 3-4 errors: mild cognitive impairment 5-7 errors: moderate cognitive impairment 8-10 errors: severe cognitive impairment

*Allow one more error for a subject with only a grade school education. Allow one less error for a subject with education beyond high school.

Source: Pfeiffer, E. (1975). A short portable mental status questionnaire for the assessment of organic brain deficit in elderly patients. Journal of American Geriatrics Society. 23, 433-41.

Exclusion criteria:

1. Inability to provide informed consent, including participation in a consent call conducted via Zoom with the study team during business hours (8:00 a.m. to 5:00 p.m. Central Time (Chicago)).
2. Participation in another research study investigating an intervention (treatments, medications, diet, or exercise). Participation in observation-only studies are not excluded.
3. Currently following a modified Paleolithic, low-fat nutrient-dense vegetarian, or Mediterranean diet with 75% OR greater reported compliance.
4. Any diagnosis or condition that is contraindicated from starting a gentle exercise program (ex. poorly controlled diseases of the heart, kidney, or liver in the prior 12 months, or severe psychiatric disease, e.g., schizophrenia, making adherence to study procedures difficult.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Modified Fatigue Impact Scale (MFIS) | Day 0 to Month 3
  Change in MFIS survey questions, scores range from 0-84, lower score is better.
Modified Fatigue Impact Scale (MFIS) | Day 0 to Month 6
  Change in MFIS survey questions, scores range from 0-84, lower score is better.
Fatigue Severity Scale (FFS) | Day 0 to Month 3
  Change in FSS survey questions, scores range from 1-63, lower score is better.
Fatigue Severity Scale (FFS) | Day 0 to Month 6
  Change in FSS survey questions, scores range from 1-63, lower score is better.
Short form 36 (SF 36) | Day 0 to Month 3
  Change in (SF 36) survey questions mean scores, range 0-100, higher number is better
Short form 36 (SF 36) | Day 0 to Month 6
  Change in (SF 36) survey questions mean scores, range 0-100, higher number is better
Rapid 3 | Day 0 to Month 3
  Change in Rapid 3 survey questions mean scores, range 0-30, lower number is better
Rapid 3 | Day 0 to Month 6
  Change in Rapid 3 survey questions mean scores, range 0-30, lower number is better

SECONDARY OUTCOMES:
Mediterranean and Paleo Diet Screener | Baseline
  Mediterranean and Paleo Diet Screener questions, scores range 0-14, higher is better
Mediterranean and Paleo Diet Screener | Month 3
  Mediterranean and Paleo Diet Screener questions, scores range 0-14, higher is better
Mediterranean and Paleo Diet Screener | Month 6
  Mediterranean and Paleo Diet Screener questions, scores range 0-14, higher is better
Hospital Anxiety and Depression Scale (HADS) | Day 0 to Month 3
  Change in HADS survey questions, scores range from 0-42, lower score is better.
Hospital Anxiety and Depression Scale (HADS) | Day 0 to Month 6
  Change in HADS survey questions, scores range from 0-42, lower score is better.
Multi-Dimensional Health Assessment Questionnaire (MDHAQ) | Day 3 to Month 3
  Change in MDHAQ survey questions, scores range from 0 to 40, lower is better
Multi-Dimensional Health Assessment Questionnaire (MDHAQ) | Day 3 to Month 6
  Change in MDHAQ survey questions, scores range from 0 to 40, lower is better

CONTACTS AND LOCATIONS:
Overall Officials: Terry L Wahls, MD, Other, Principal Investigator — University of Iowa
Locations (1):
- Univeristy of Iowa, Iowa City, Iowa, United States

REFERENCES:
- [Background] Sandikci SC, Ozbalkan Z. Fatigue in rheumatic diseases. Eur J Rheumatol. 2015 Sep;2(3):109-113. doi: 10.5152/eurjrheum.2015.0029. Epub 2015 Sep 1. PMID 27708942
- [Background] Wolfe F, Hawley DJ, Wilson K. The prevalence and meaning of fatigue in rheumatic disease. J Rheumatol. 1996 Aug;23(8):1407-17. PMID 8856621
- [Background] Nikolaus S, Bode C, Taal E, van de Laar MA. Fatigue and factors related to fatigue in rheumatoid arthritis: a systematic review. Arthritis Care Res (Hoboken). 2013 Jul;65(7):1128-46. doi: 10.1002/acr.21949. PMID 23335492
- [Background] Omdal R, Mellgren SI, Koldingsnes W, Jacobsen EA, Husby G. Fatigue in patients with systemic lupus erythematosus: lack of associations to serum cytokines, antiphospholipid antibodies, or other disease characteristics. J Rheumatol. 2002 Mar;29(3):482-6. PMID 11908560
- [Background] Miller FW. The increasing prevalence of autoimmunity and autoimmune diseases: an urgent call to action for improved understanding, diagnosis, treatment, and prevention. Curr Opin Immunol. 2023 Feb;80:102266. doi: 10.1016/j.coi.2022.102266. Epub 2022 Nov 26. PMID 36446151
- [Background] Dean C, Parks S, Titcomb TJ, Arthofer A, Meirick P, Grogan N, Ehlinger MA, Bisht B, Fox SS, Daack-Hirsch S, Snetselaar LG, Wahls TL. Facilitators of and Barriers to Adherence to Dietary Interventions Perceived by Women With Multiple Sclerosis and Their Support Persons. Int J MS Care. 2022 Sep-Oct;24(5):235-241. doi: 10.7224/1537-2073.2021-051. Epub 2022 May 26. PMID 36090239